

# NON-INTERVENTIONAL (NI) STUDY PROTOCOL

# **Study Information**

| Title | Novel Hormonal Therapy (NHT) for Treating Patients with<br>Metastatic Castration-Sensitive Prostate Cancer (mCSPC): An<br>Analysis of National Veterans Affairs Health Care Network<br>Data |
|---|---|
| Protocol number | C3431052 |
| Protocol version identifier | 1.0 |
| Date | 06 November 2023 |
| Active substance | Enzalutamide |
| Medicinal product | Xtandi |
| Research question and objectives | 06 November 2023<br>Enzalutamide |

| | CCI |
|---|---|
| | 4. Describe time to deep prostate-specific antigen (PSA) response and time to undetectable PSA overall |
| | 5. Describe time to progression overall CCI |
| | 6. Describe the distribution of next therapy regimens overall |
| Author | PPD , MA |
| | PPD |
| | Pfizer Inc. |
| | PPD |

This document contains confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

| 1. TABLE OF CONTENTS 3 2. LIST OF ABBREVIATIONS 5 3. RESPONSIBLE PARTIES 7 4. ABSTRACT 8 5. AMENDMENTS AND UPDATES 11 6. MILESTONES 12 7. RATIONALE AND BACKGROUND 13 8. RESEARCH QUESTION AND OBJECTIVES 13 9. RESEARCH METHODS 14 9.1. Study Design 14 9.2. Setting 14 9.2. Setting 17 9.3. Variables 17 9.4. Data Sources 22 9.5. Study Size 22 9.6. Data Management 22 9.7. Data Analysis for Primary Objective: Describe TTNT among patients with mCSPC who initiated NHT in 1L 22 9.7.2. Data Analysis for Secondary Objective: Describe TTNT among patients with mCSPC who initiated NHT in 1L 23 9.7.3. Data Analysis for Exploratory Objectives 23 9.7.3.1. Data Analysis for Exploratory Objectives 23 9.7.3.2. Data Analysis for Exploratory Objective 1: Describe patient baseline characteristics overall 23 9.7.3.3. Data Analysis for Exploratory Objective 4: Describe time to deep prostate-specific antigen (PSA) response and time to undetectable PSA overall 24 <th>1. TABLE OF CONTENTS</th> <th></th> | 1. TABLE OF CONTENTS | |
|---|---|---|
| 3. RESPONSIBLE PARTIES | 1. TABLE OF CONTENTS | 3 |
| 4. ABSTRACT | 2. LIST OF ABBREVIATIONS | 5 |
| 5. AMENDMENTS AND UPDATES | 3. RESPONSIBLE PARTIES | 7 |
| 6. MILESTONES | 4. ABSTRACT | 8 |
| 7. RATIONALE AND BACKGROUND 13 8. RESEARCH QUESTION AND OBJECTIVES 13 9. RESEARCH METHODS 14 9.1. Study Design 14 9.2. Setting 14 9.2.1. Inclusion Criteria 15 9.2.2. Exclusion Criteria 17 9.3. Variables 17 9.4. Data Sources 22 9.5. Study Size 22 9.6. Data Management 22 9.7. Data Analysis 22 9.7.1. Data Analysis for Primary Objective: Describe TTNT among patients with mCSPC who initiated NHT in 1L 22 9.7.2. Data Analysis for Secondary Objective: Describe TTNT among patients with mCSPC who initiated NHT in 1L 23 9.7.3. Data Analysis for Exploratory Objectives 23 9.7.3.1. Data Analysis for Exploratory Objective 1: Describe patient baseline characteristics overall 23 9.7.3.3. Data Analysis for Exploratory Objective 4: Describe time to deep prostate-specific antigen (PSA) response and time to undetectable PSA overall | 5. AMENDMENTS AND UPDATES | 11 |
| 8. RESEARCH QUESTION AND OBJECTIVES | 6. MILESTONES | 12 |
| 9. RESEARCH METHODS | 7. RATIONALE AND BACKGROUND | 13 |
| 9.1. Study Design | 8. RESEARCH QUESTION AND OBJECTIVES | 13 |
| 9.2. Setting | 9. RESEARCH METHODS | 14 |
| 9.2.1. Inclusion Criteria | 9.1. Study Design | 14 |
| 9.2.2. Exclusion Criteria | 9.2. Setting. | 14 |
| 9.3. Variables | 9.2.1. Inclusion Criteria | 15 |
| 9.4. Data Sources | 9.2.2. Exclusion Criteria | 17 |
| 9.5. Study Size | 9.3. Variables | 17 |
| 9.6. Data Management | 9.4. Data Sources | 22 |
| 9.7. Data Analysis | 9.5. Study Size | 22 |
| 9.7.1. Data Analysis for Primary Objective: Describe TTNT among patients with mCSPC who initiated NHT in 1L | 9.6. Data Management | 22 |
| patients with mCSPC who initiated NHT in 1L | 9.7. Data Analysis | 22 |
| patients with mCSPC who initiated NHT in 1L | | 22 |
| 9.7.3.1. Data Analysis for Exploratory Objective 1: Describe patient baseline characteristics overall 23 9.7.3.3. Data Analysis for Exploratory Objective 4: Describe time to deep prostate-specific antigen (PSA) response and time to undetectable PSA overall | | .23 |
| patient baseline characteristics overall 23 CCI 23 9.7.3.3. Data Analysis for Exploratory Objective 4: Describe time to deep prostate-specific antigen (PSA) response and time to undetectable PSA overall | 9.7.3. Data Analysis for Exploratory Objectives | 23 |
| 9.7.3.3. Data Analysis for Exploratory Objective 4: Describe time to deep prostate-specific antigen (PSA) response and time to undetectable PSA overall | | |
| 9.7.3.3. Data Analysis for Exploratory Objective 4: Describe time to deep prostate-specific antigen (PSA) response and time to undetectable PSA overall | | 23 |
| to deep prostate-specific antigen (PSA) response and time to undetectable PSA overall | | .23 |
| | to deep prostate-specific antigen (PSA) response and time to undetectable PSA overall | 24 |

| 9.7.3.4. Data Analysis for Exploratory Objective 5: Describe time to progression overall CCI | 24 |
|---|---|
| 9.7.3.5. Data Analysis for Exploratory Objective 6: Describe the distribution of next therapy regimens overall | 24 |
| 9.8. Quality Control | 25 |
| 9.9. Limitations of the Research Methods | 25 |
| 9.10. Other Aspects | 25 |
| 10. PROTECTION OF HUMAN PARTICIPANTS | 26 |
| 10.1. Patient Information | 26 |
| 10.2. Patient Consent | 26 |
| 10.3. Institutional Review Board (IRB)/ Ethics Committee (EC) | 26 |
| 10.4. Ethical Conduct of the Study | 26 |
| 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 26 |
| 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | 26 |
| 13. REFERENCES | 27 |
| 14. LIST OF TABLES | 29 |
| 15. LIST OF FIGURES | 29 |
| ANNEX 1. LIST OF STANDALONE DOCUMENTS | 29 |
| ANNEX 2. ADDITIONAL INFORMATION | 30 |

# 2. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| ABI | abiraterone acetate |
| ADT | Androgen Deprivation Therapy |
| AE | adverse event |
| APA | apalutamide |
| CCI | Charlson Comorbidity Index |
| CDW | Corporate Data Warehouse |
| CI | confidence interval |
| CRPC | castration-resistant prostate cancer |
| CSPC | castration-sensitive prostate cancer |
| DOT | duration of treatment |
| EC | Ethics Committee |
| ENZ | enzalutamide |
| FDA | United States Food and Drug Administration |
| ICD-10-CM | International Classification of Diseases, 10th<br>Revision, Clinical Modification |
| IPTW | Inverse probability treatment weighting |
| IRB | Institutional Review Board |
| KM | Kaplan-Meier |
| mCRPC | metastatic CRPC |
| mCSPC | metastatic CSPC |
| NCI | National Cancer Institute |

| Abbreviation | Definition |
|--------------|-------------------------------------------------|
| NHT | Novel Hormonal Therapy |
| NSAA | non-steroidal anti-androgen |
| PC | prostate cancer |
| РН | proportional hazards |
| PSA | prostate-specific antigen |
| PFS | progression-free survival |
| SAS | Statistical Analysis System |
| SLVHCS | Southeast Louisiana Veterans Health Care System |
| SMD | Standardized Mean Difference |
| TTNT | time to next therapy |
| VA | Veterans' Affairs |
| VHA | Veterans' Health Administration |

# 3. RESPONSIBLE PARTIES

# Principal Investigator(s) of the Protocol

| Name, Degree(s) | Job Title | Affiliation | Address |
|---|---|---|---|
| Jasmina Ivanova, MA | Senior Director, Value & Evidence – Xtandi Patient & Health Impact | Pfizer Inc. | 66 Hudson Blvd.<br>New York New York 10001 |
| Dave Russell, MD | Senior Director, Global<br>Medical Affairs, Xtandi<br>Lead | Pfizer Inc. | 66 Hudson Blvd.<br>New York New York 10001 |
| Maelys Touya, PharmD, MSc | Director, HEOR<br>Oncology | Astellas Pharma<br>US, Inc. | 2375 Waterview Drive<br>Northbrook, IL 60062 |
| Hongbo Yang, PhD, MS | Vice President | Analysis Group | 111 Huntington Ave<br>14 <sup>th</sup> Floor<br>Boston, MA 02199 |
| Wei Gao, PhD, MS | Vice President | Analysis Group | 111 Huntington Ave<br>14 <sup>th</sup> Floor<br>Boston, MA 02199 |

#### 4. ABSTRACT

**Title:** Novel Hormonal Therapy (NHT) for Treating Patients with Metastatic Castration-Sensitive Prostate Cancer (mCSPC): An Analysis of National Veterans Affairs Health Care Network Data

Version: 1.0

Date of Protocol: 06 November 2023

**Author:** 

PPD

Rationale and Background: Prostate cancer is the most common cancer and the second leading cause of cancer death among men in the United States. While the long-term outlook is positive for early-stage prostate cancer, survival rates drastically decrease once the disease has spread beyond the prostate gland. Metastatic castration-sensitive prostate cancer (mCSPC) is form of metastatic prostate cancer among men who have never received or are sensitive to androgen deprivation therapy (ADT). Conventional therapy for mCSPC has been ADT, however, mCSPC treated with ADT might eventually transition to castration-resistant prostate cancer (CRPC) stage with a median survival of approximately 3 years. Upfront intensified treatment with NHTs, including abiraterone acetate (ABI), apalutamide (APA), and enzalutamide (ENZ), added to a backbone of ADT, has substantially improved survival in clinical trials. Due to relatively recent approval of NHTs in mCSPC there is limited information on real-world duration of treatment and time to next treatment with these therapies. The current study proposes to use the Veterans Health Administration (VHA) database to describe outcomes of patients with NHT use in mCSPC.

**Objectives:** The study objectives include:

- **Primary objective:** Describe duration of therapy (DOT) among patients with mCSPC who initiated NHT in the first line (1L)
- **Secondary objective:** Describe time to next therapy (TTNT) among patients with mCSPC who initiated NHT in 1L.
- Exploratory objectives:

| 1. | Describe patient baseline characteristics overall CC |
|----|------------------------------------------------------|
| CC | CCI |

- 4. Describe time to deep prostate-specific antigen (PSA) response and time to undetectable PSA overall CCI
- 5. Describe time to progression overall
- 6. Describe the distribution of next therapy regimens overall

**Study Design:** This is a retrospective, observational study using the VHA data. Patients with mCSPC who initiated NHT in 1L during January 2020 – December 2022 will be selected based on diagnosis history, treatment history, PSA measurements, age, and continuous enrollment.

Patients will be required to have 365 days of continuous enrollment in the National Veterans' Affairs (VA) Health Care Network prior to their index date, during which baseline characteristics will be assessed. The follow-up period will be defined as the time from the index date to the end of continuous enrollment, the end of the data availability, or death, whichever comes first. During the follow-up period, the outcome measures (ie, DOT, TTNT, time to deep PSA response, time to undetectable PSA, time to progression, and the distribution of next treatment) will be assessed.

**Population:** The population for the primary and secondary objectives will consist of patients with mCSPC who initiated NHT in 1L and who meet all the sample selection criteria.

**Variables**: Baseline demographic and clinical characteristics will include age, race, geographic regions, index year, treatment history, diagnosis history, prognostic variables, Charlson Comorbidity Index score, and individual comorbidities. Outcomes will include DOT, TTNT, time to deep PSA response, time to undetectable PSA, and time to progression.

**Data Sources:** VHA Medical Statistical Analysis System datasets.

**Study Size:** All eligible patients available for the analysis will be included.

**Data Analysis:** In the primary and secondary analyses, DOT and TTNT will be described in the overall sample of patients with mCSPC who initiated 1L NHT using Kaplan-Meier (KM) analysis. The number at risk table and the median time to event and its 95% confidence interval will be reported. In the exploratory analyses, patient baseline characteristics will be described in the overall sample Means, standard deviations, medians, and interquartile range will be e ous variables; counts and percentages will be estimated for categorical variables.

KM analysis will be conducted to describe time to deep PSA response, time to

Data analysis will be executed using statistical software SAS version 9.4 (Cary, NC).

# 5. AMENDMENTS AND UPDATES

None.

# 6. MILESTONES

| Milestone | Planned Date |
|--------------------------|------------------|
| Start of data collection | 21 November 2023 |
| End of data collection | 31 October 2024 |
| Final study report | 31 December 2024 |

#### 7. RATIONALE AND BACKGROUND

Prostate cancer is the most common cancer and the second leading cause of cancer death among men in the United States. The National Cancer Institute estimates that in 2022 there will be 268,490 new cases of prostate cancer (PC) and 34,500 deaths due to PC.8 While the long-term outlook is positive for early-stage prostate cancer, survival rates drastically decrease once the disease has spread beyond the prostate gland.9

Metastatic castration-sensitive prostate cancer (mCSPC) is form of metastatic prostate cancer among men who have never received or are sensitive to ADT.<sup>5</sup> Conventional therapy for mCSPC has been ADT, however, mCSPC treated with ADT might eventually transition to CRPC stage with a median survival of approximately 3 years.<sup>11</sup>

Several NHTs have been approved for treatment in mCSPC together with ADT. ABI and ENZ were initially approved by the United States Food and Drug Administration (FDA) for metastatic CRPC patients with prior chemotherapy in April 2011 and August 2012, respectively, and for chemotherapy-naïve patients in December 2012 and September 2014, respectively. ABI was later approved in February 2018, followed by ENZ in December 2019, for the treatment of mCSPC. <sup>1,2</sup> One of the most recent NHTs, apalutamide (APA) was approved by the FDA in September 2019 for patients with mCSPC.<sup>3</sup>

Upfront intensified treatment with NHTs in mCSPC, including ABI, APA, and ENZ, added to a backbone of ADT, has substantially improved survival.<sup>4,6,10</sup> With the rapidly expanding treatment landscape, there have been limited studies describing clinical outcomes with NHTs in mCSPC.

The current study proposes to use the VHA database to describe outcomes of patients with NHT use in in mCSPC.

### 8. RESEARCH OUESTION AND OBJECTIVES

The main research question is to identify men with mCSPC from the VHA database who were treated with NHT, including ABI, APA, and ENZ, in the 1L setting and describe clinical outcomes of interest.

More specifically, the study objectives include:

- **Primary objective:** Describe DOT among patients with mCSPC who initiated NHT in 1L
- **Secondary objective:** Describe TTNT among patients with mCSPC who initiated NHT in 1L

# • Exploratory objectives:



### 9. RESEARCH METHODS

## 9.1. Study Design

This is a retrospective, observational study using the VHA data. Patients with mCSPC who initiated NHT in 1L during January 2020 – December 2022 will be selected based on diagnosis history, treatment history, PSA measurements, age, and continuous enrollment.

6. Describe the distribution of next therapy regimens overall

Patients will be required to have one year of continuous enrollment in the National VA Health Care Network prior to their index date, during which patient baseline characteristics will be assessed. The time period (January 2020 – December 2022) to identify NHT initiation reflects the recency of NHT approvals, and the baseline period allows us to capture any potential comorbidities and characteristics that may be confounders to the outcomes. The follow-up period will be defined as the time from the index date to the end of continuous enrollment, the end of the data availability, or death, whichever comes first. During the follow-up period, the outcome measures (ie, DOT, TTNT, time to deep PSA response, time to undetectable PSA, time to progression, and the distribution of next treatment) will be assessed. The follow-up period is chosen to maximally capture any potential outcomes among patients with mCSPC who initiated NHT in 1L.

# 9.2. Setting

The study population will include patients with mCSPC who initiated NHT in 1L in the VHA database. Inclusion and exclusion criteria are specified below.

#### 9.2.1. Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

- Males.
- Have at least one claim with a diagnosis code of PC (PC; ICD-10-CM code C61).
- Have documented secondary metastasis codes on or after the initial PC diagnosis (ICD-10 codes C77, C78, C79, C7B).
- Have initiated ABI, APA, or ENZ (1) during the index window of January 2020 –
  December 2022, and (2) within 90 days prior to or any time after the first claim for
  metastatic disease. The initiation of date of ABI, APA, or ENZ will be defined as the
  index date.
  - Index window of January 2020 December 2022 is selected, as during this period all NHTs were approved for mCSPC, which will help remove early initiator bias (eg, when a product/class of products became available, patients with severe diseases tend to try first). Table 1 lists the approval dates for when each NHT was approved for treating mCSPC.

Table 1. FDA Approval Dates for NHTs in mCSPC

| ABI | 07 February 2018 |
|-----|-------------------|
| APA | 17 September 2019 |
| ENZ | 16 December 2019 |

- At least 18 years old at the index date.
- Have continuous enrollment for at least 365 days before the index date.
- Have evidence to be castration sensitive AND have no evidence to be castration resistant. This is tentatively defined as:

#### Evidence to be castration sensitive:

- No prior surgical castration (ie, bilateral orchiectomy, Appendix Table 1) any time prior to the index date or no medical castration (ie, degarelix, relugolix, goserelin, histrelin, leuprolide, and triptorelin; ≥8 weeks of continuous use; Appendix Table 1) within -90 to -365 days prior to the index date, OR
- Presence of ICD-10-CM diagnosis code indicating hormone sensitive malignancy status (ie, Z19.1, which was introduced on 01 October 2016) within 90 days before the index date

### *No evidence to be castration resistant:*

- No evidence of castration resistance any time prior to the index date. Evidence of castration resistance is defined by the following:
  - ICD-10-CM diagnosis code indicating hormone resistance (Z19.2), OR
  - A rise in PSA from the nadir by ≥2 ng/mL after castration (nadir is defined as the lowest PSA since surgical or medical castration and before the index date)
  - Patients with other PC treatment including NHT, non-steroidal antiandrogen (NSAA), chemotherapy, immunotherapy, radium 223, lutetium Lu 177 vipivotide tetraxetan, ketoconazole, niraparib, olaparib, rucaparib, or talazoparib at any time prior to the index date

Figure 1. Study Schema



### 9.2.2. Exclusion Criteria

Patients meeting any of the following criteria will not be included in the study:

- Patients with any other primary cancer (excluding non-melanoma skin cancer) prior to the index date
- Participation in clinical trial during the 30 days prior to the index date



### 9.3. Variables

Table 2. Baseline Demographics and Clinical Characteristics

| Variable | Operational Definition |
|---|---|
| Baseline period | The baseline period will be defined as 365 days prior to the index date. |
| Age | Age will be defined as of the index date and retained in the dataset as a continuous variable and a categorical variable: 18-49, 50-59, 60-69, 70-79, and ≥80 years old. |
| Race | Proportion of patients that were Hispanic, non-Hispanic white, black, other, and unknown races will be evaluated. |

| Variable | Operational Definition |
|---|---|
| Geographic regions | Proportion of patients that lived in Northeast, Midwest, South and West areas. |
| Index year | Variable will be created for the index calendar year (from 2020 to 2022). |
| Treatment history | Proportion of patients who had radical prostatectomy, external radiotherapy, chronic corticosteroid use, hormone therapy, bone protective agents, and pain medication prescribed in the baseline period will be evaluated. |
| Time from Metastatic<br>Diagnosis Date to Index<br>Date | Time from the first observed metastatic date in the data to the index date will be evaluated. |
| Time from PC Diagnosis<br>Date to Index Date | Time from the first observed PC date in the data to the index date will be evaluated. |
| Site of Metastasis | Flags will be created for patients that had a metastatic diagnosis at the following sites: bone only, bone and node only, node only, viscera and other. |
| PSA Value | Baseline PSA value (if available) will be defined as the PSA value closest to the index date within 180 days prior to index date. |
| Hemoglobin Value | Baseline hemoglobin value (if available) will be defined as the value closest to the index date within 180 days prior to index date. |
| Alkaline Phosphatase<br>Value | Baseline alkaline phosphatase value (if available) will be defined as the value closest to the index date within 180 days prior to index date. |
| Modified National Cancer<br>Institute (NCI) Charlson<br>Comorbidity Index (CCI) | The NCI CCI score excluding cancer will be calculated during the baseline period. |
| Acute Coronary Syndrome | A binary variable (yes/no) will be created for patients with claims for acute coronary syndrome during the baseline period. |
| Angina Pectoris | A binary variable (yes/no) will be created for patients with claims for angina pectoris during the baseline period. |

| Variable | Operational Definition |
|---|---|
| Arrhythmia | A binary variable (yes/no) will be created for patients with claims for arrhythmia during the baseline period. |
| Chronic Obstructive<br>Pulmonary Disease | A binary variable (yes/no) will be created for patients with claims for chronic obstructive pulmonary disease during the baseline period. |
| Congestive Heart Failure | A binary variable (yes/no) will be created for patients with claims for congestive heart failure during the baseline period. |
| Diabetes | A binary variable (yes/no) will be created for patients with claims for diabetes (types 1 and 2) during the baseline period. |
| Hyperlipidemia | A binary variable (yes/no) will be created for patients with claims for hyperlipidemia during the baseline period. |
| Hypertension | A binary variable (yes/no) will be created for patients with claims for hypertension during the baseline period. |
| Inflammatory Bowel<br>Disease | A binary variable (yes/no) will be created for patients with claims for inflammatory bowel disease (ulcerative colitis, Crohn's disease) during the baseline period. |
| Lower-extremity Arterial<br>Occlusive Disease | A binary variable (yes/no) will be created for patients with claims for low-extremity arterial occlusive disease during the baseline period. |
| Myocardial Infarction | A binary variable (yes/no) will be created for patients with claims for myocardial infraction during the baseline period. |
| Stroke | A binary variable (yes/no) will be created for patients with claims for stroke during the baseline period. |

Table 3. Outcomes During the Follow-up Period

| Variable | Operational Definition |
|---|---|
| Follow-up period | The follow-up period will be defined as the time from the index date to the end of continuous enrollment, the end of the data availability, or death, whichever comes first. |
| DOT | Duration of therapy will be defined as the time from the index date to the date of NHT discontinuation for any reason. Discontinuation of the current NHT will be defined as a treatment gap of at least 90 days (the last day with days supply before the gap as discontinuation date), the initiation of a new therapy, or death, whichever comes first. Initiation of a new therapy will be defined by switching to a different NHT, switching to or augmentation with NSAA, chemotherapy, immunotherapy, radium 223, lutetium Lu 177 vipivotide tetraxetan, ketoconazole, niraparib, olaparib, rucaparib, or talazoparib. Patients who do not experience discontinuation will be censored at the end of data availability. |
| TTNT | Time to next therapy will be defined as the time from the index date to the initiation date of a new therapy (see the definition of a new therapy above). Patients who do not initiate a new therapy will be censored at the end of data availability or death, whichever comes first. |
| Next therapy regimen | The next therapy regimen will include all therapies noted below initiated within 28 days of the start of the new therapy (different NHT, switching to or augmentation with NSAA, chemotherapy, immunotherapy, radium 223, lutetium Lu 177 vipivotide tetraxetan, ketoconazole, niraparib, olaparib, rucaparib, or talazoparib). |
| PSA assessment and PSA response description | <ul> <li>The following will be described for patients with a baseline and at least one post baseline PSA value:</li> <li>The distribution of the number of post baseline PSA assessments</li> <li>PSA nadir (lowest post-baseline value)</li> <li>Number and proportion of patients with deep PSA</li> </ul> |
| | • Number and proportion of patients with deep PSA response (≥ 90% decrease in a post-index PSA value |

| Variable | Operational Definition |
|---|---|
| | from the baseline PSA value) any time during follow-up • Number and proportion of patients with undetectable PSA value post baseline (using different thresholds): |
| | <ul><li>&lt;0.2 ng/mL</li><li>&lt;0.1 ng/mL</li></ul> |
| | • <0.01 ng/mL |
| Time to deep PSA response | Time to deep PSA response will be calculated among patients who have baseline PSA value and at least one PSA value after the index date. Time to deep PSA response will be defined as the time from the index date to the date of deep PSA response. Deep PSA response will be defined as ≥90% decrease in a post-index PSA value from the baseline PSA value. Patients who do not experience deep PSA response will be censored at the end of last available PSA assessment. |
| Time to undetectable PSA | Time to undetectable PSA will be calculated among patients who have baseline PSA value and at least one PSA value after the index date. Time to undetectable PSA will be defined as the time from the index date to the first evidence of undetectable PSA. Undetectable PSA may be defined using different thresholds (eg, <0.2 ng/mL). Patients who do not have undetectable PSA post index will be censored at the end of last available PSA assessment. |
| Time to progression | Time to progression will be defined as the time from the index date to the first evidence of disease progression. Progression will be defined as PSA progression, initiation of a new therapy, or death, whichever comes first. PSA progression will be defined as an increase of ≥25% and an absolute increase of ≥2ng/mL in PSA from the nadir value post-index. Patients who do not experience disease progression will be censored at the end of data availability. |

#### 9.4. Data Sources

Data from the National VA Health Care Network will be used for this study. This network is the U.S.'s largest integrated health care system with over 1,700 sites of care, serving approximately 8.76 million veterans each year. The VA Health System Corporate Data Warehouse (CDW) includes all medical encounter information in the VA, comprised of medical centers, community-based outpatient clinics, community-living centers, veteran centers, and domiciliaries. The VA CDW stores data in separate databases, one for each type of clinical information - inpatient medication, inpatient laboratory, inpatient admission, outpatient medication, outpatient visits, etc. The databases provide demographic information and contain comprehensive services, including primary care, specialty care, inpatient care, rehabilitation, long-term care, home care, and other services, to military veterans. The database also includes date of death. The date of death is extracted from the VA electronic health record systems and verified by official sources, including VA facilities, death certificates, and National Cemetery Administration. Information on CDW, including date of death, is updated on a daily base. Cause of death is not available on CDW.

### 9.5. Study Size

As no priori hypotheses are specified, sample size calculations are not applicable. The number of patients eligible for the study will be determined in accordance with the sample selection conducted per the criteria described in Section 9.2.

# 9.6. Data Management

A clean, patient-level dataset will be generated for use throughout the study. This process will entail basic exploratory checks to ensure data integrity; cleaning and reformatting the raw data as needed; and creating variables for all key study measures, including patient characteristics, treatment start and end dates, and classification of treatments and medication. All data will be stored and maintained on National VA Health Care Network and accessed over Southeast Louisiana Veterans Health Care System (SLVHCS) at Tulane University. The data will be made accessible only to individuals working on the current study. No attempt will be made to identify individual patients, hospitals, or physicians. Analyses will be conducted using SAS 9.4 (SAS Institute, Cary NC).

#### 9.7. Data Analysis

# 9.7.1. Data Analysis for Primary Objective: Describe TTNT among patients with mCSPC who initiated NHT in 1L

DOT, as defined in Table 3, will be summarized among the overall sample of patients with mCSPC who initiated NHT in 1L. Kaplan-Meier (KM) analysis will be used to describe DOT, and patients who do not experience treatment discontinuation will be censored at the end of data availability. The number of patients at risk and the number and proportion of individuals experiencing discontinuation during the follow-up period (eg, annually or every 6 months) will be reported. The median DOT and corresponding 95% CI will be reported.

# 9.7.2. Data Analysis for Secondary Objective: Describe TTNT among patients with mCSPC who initiated NHT in 1L

TTNT, as defined in Table 3, will be summarized among the overall sample of patients with mCSPC who initiated NHT in 1L. KM analysis will be used to describe TTNT, and patients who do not initiate a new therapy will be censored at the end of data availability. The number of patients at risk and the number and proportion of individuals initiating a new therapy during the follow-up period (eg, annually or every 6 months) will be reported. The median TTNT and corresponding 95% CI will be reported.

# 9.7.3. Data Analysis for Exploratory Objectives





# 9.7.3.4. Data Analysis for Exploratory Objective 5: Describe time to progression overall

Time to progression, as defined in Table 3, will be summarized in the overall sample of patients with mCSPC who initiated 1L NHT

# 9.7.3.5. Data Analysis for Exploratory Objective 6: Describe the distribution of next therapy regimens overall

The number and proportion of patients who initiated a new therapy following the index NHT will be estimated in the overall sample CCI

Among those who initiated a new therapy, the number and proportion of patients who received different type of regimen for first subsequent therapy will be described. A noted in Table 3, the next therapy regiment will include all therapies noted below initiated within 28 days of the start of the new therapy (different NHT, switching to or augmentation with NSAA, chemotherapy, immunotherapy, radium 223, lutetium Lu 177 vipivotide tetraxetan, ketoconazole, niraparib, olaparib, rucaparib, or talazoparib).

# 9.8. Quality Control

Best practice guidelines will be followed to ensure project quality, including structured organization of project materials (eg, data extracts, statistical software programs, output tables) and standard internal audit process. The audit process both confirms the validity of the analytical approach and ensures that all programs and results are accurate.

### 9.9. Limitations of the Research Methods

The analyses conducted as part of this study are subject to the following limitations, which will be addressed in any write-up of the study:

- As this study will be conducted among veterans, its findings may not be generalizable to other populations.
- Also, as we are pulling VA only data, we are not able to capture care that occurs
  outside the VA which could lead to missing data and misclassification of disease
  states and treatment groups.
- There are no specific diagnosis codes for CSPC. Assumptions will be made to select patients with CSPC based on clinical input.
- Certain assumptions will be made in order to depict treatment patterns for determining TTNT. However, the definition of treatment patterns will nevertheless be subject to assumptions that may not match up to the prescribing physicians' intent.
- Data are subject to inaccuracies in coding of diagnoses. The presence of a diagnosis code in the data does not necessarily mean the presence of disease. The disease may be incorrectly coded or the code was included as a rule-out criterion.
- The presence of a prescription does not necessarily mean the medication was used as prescribed. In addition, prescriptions filled over the counter or provided as samples by the physician are not included in the data.
- Regression models cannot account for unmeasured factors.

### 9.10. Other Aspects

Not applicable.

#### 10. PROTECTION OF HUMAN PARTICIPANTS

#### 10.1. Patient Information

This study involves data that exist in deidentified/anonymized structured format and contain no patient personal information.

### 10.2. Patient Consent

As this study involves deidentified/anonymized structured data, which according to applicable legal requirements do not contain data subject to privacy laws, obtaining informed consent from patients by Pfizer is not required.

# 10.3. Institutional Review Board (IRB)/ Ethics Committee (EC)

This protocol, and any subsequent modifications, will be reviewed and approved by the SLVHCS IRB prior to implementation.

# 10.4. Ethical Conduct of the Study

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value, and rigor and follow generally accepted research practices described in Guidelines for Good Pharmacoepidemiology Practices (GPP). Public Policy Committee, International Society of Pharmacoepidemiology. Pharmacoepidemiology and Drug Safety 2015; 25:2-10. https://onlinelibrary.wiley.com/doi/full/10.1002/pds.3891.

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

This study involves data that exist as structured data by the time of study start. In these data sources, individual patient data are not retrieved or validated, and it is not possible to link (ie, identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (ie, identifiable patient, identifiable reporter, a suspect product, and event) cannot be met.

### 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

Based on the analysis results and discussions with Pfizer, a study report summarizing the background, objectives, methods, results, and conclusion of the study will be prepared. The study report may be disseminated within Pfizer but is not expected to be externally communicated.

In the event of any prohibition or restriction imposed (eg, clinical hold) by an applicable competent authority in any area of the world, or if the party responsible for collecting data from the participant is aware of any new information which might influence the evaluation of the benefits and risks of a Pfizer product, Pfizer should be informed immediately.

### 13. REFERENCES

- US Food and Drug Administration. FDA approves abiraterone acetate in combination
  with prednisone for high-risk metastatic castration-sensitive prostate cancer 2018
  [Available from: https://www.fda.gov/drugs/resources-information-approved-drugs/fdaapproves-abiraterone-acetate-combination-prednisone-high-risk-metastatic-castrationsensitive].
- 2. US Food and Drug Administration. FDA approves enzalutamide for metastatic castration-sensitive prostate cancer 2019 [Available from: https://www.fda.gov/drugs/resources-information-approved-drugs/fda-approves-enzalutamide-metastatic-castration-sensitive-prostate-cancer].
- 3. US Food and Drug Administration. FDA approves apalutamide for metastatic castration-sensitive prostate cancer 2019 [Available from: https://www.fda.gov/drugs/resources-information-approved-drugs/fda-approves-apalutamide-metastatic-castration-sensitive-prostate-cancer].
- 4. Chi KN, Agarwal N, Bjartell A, Chung BH, Pereira de Santana Gomes AJ, Given R, et al. Apalutamide for Metastatic, Castration-Sensitive Prostate Cancer. N Engl J Med. 2019;381(1):13-24.
- 5. Damodaran S, Lang JM, Jarrard DF. Targeting Metastatic Hormone Sensitive Prostate Cancer: Chemohormonal Therapy and New Combinatorial Approaches. J Urol. 2019;201(5):876-85.
- 6. Davis ID, Martin AJ, Stockler MR, Begbie S, Chi KN, Chowdhury S, et al. Enzalutamide with Standard First-Line Therapy in Metastatic Prostate Cancer. N Engl J Med. 2019;381(2):121-31.
- 7. National Cancer Institute. Prostate Cancer 2022 [Available from: https://www.cancer.gov/types/prostate].
- 8. National Cancer Institute. Cancer Stat Facts: Prostate Cancer 2022 [Available from: https://seer.cancer.gov/statfacts/html/prost.html].
- 9. National Cancer Institute. Prostate Cancer Treatment Health Professional Version 2022 [Available from: https://www.cancer.gov/types/prostate/hp/prostate-treatment-pdq].
- 10. Rydzewska LHM, Burdett S, Vale CL, Clarke NW, Fizazi K, Kheoh T, et al. Adding abiraterone to androgen deprivation therapy in men with metastatic hormone-sensitive prostate cancer: A systematic review and meta-analysis. Eur J Cancer. 2017;84:88-101.

11. Tangen CM, Hussain MH, Higano CS, Eisenberger MA, Small EJ, Wilding G, et al. Improved overall survival trends of men with newly diagnosed M1 prostate cancer: a SWOG phase III trial experience (S8494, S8894 and S9346). J Urol. 2012;188(4):1164-9.

# 14. LIST OF TABLES

- Table 1. FDA Approval Dates for NHTs in mCSPC
- Table 2. Baseline Demographics and Clinical Characteristics
- Table 3. Outcomes During the Follow-up Period

# 15. LIST OF FIGURES

Figure 1. Study Schema

# ANNEX 1. LIST OF STANDALONE DOCUMENTS

None.

# **ANNEX 2. ADDITIONAL INFORMATION**

# **Appendix Table 1. Codes for Treatments**

| Hormonal therapy | GPI | HCPCS/CPT | ICD |
|---|---|---|---|
| Androgen deprivation therapy | | | |
| Bilateral orchiectomy | | <u>CPT</u> 54520, 54522, 54530, 54535, 54690 | <u>ICD-9-CM</u><br>V45.77 |
| Identified by having at least one procedure code for bilateral orchiectomy, having unilateral procedure codes for both testicles (left and right), or having two unilateral orchiectomy | | | <u>ICD-10-CM</u><br>Z90.79 |
| procedures (location unspecified) on different dates | | | <u>ICD-9-PCS</u><br>623, 6241, 6242 |
| | | | ICD-10-PCS<br>0V590ZZ, 0V593ZZ, 0V594ZZ, 0V5B0ZZ,<br>0V5B3ZZ, 0V5B4ZZ, 0V5C0ZZ, 0V5C3ZZ,<br>0V5C4ZZ, 0VT90ZZ, 0VT94ZZ, 0VTB0ZZ,<br>0VTB4ZZ, 0VTC0ZZ, 0VTC4ZZ |
| LHRH agonists/antagonists | | | |
| Degarelix | 2140552510 | J9155 | |
| Relugolix | 21405570000320<br>24993503800320 | | |
| Goserelin | 21405005 | J9202 | |
| Histrelin | 2140500710 | J1675, J9225, J9226, S0133 | |
| Leuprolide | 21405010 | J1950, J9217, J9218, J9219, Q0057 | |
| Triptorelin | 21405050 | J3315 | |
| Novel hormonal therapy | | | |
| Apalutamide | 2140241000 | | |
| Abiraterone | 2140601020 | | |
| Darolutamide | 2140242500 | | |
| Enzalutamide | 2140243000 | | |
| Non-steroidal anti-androgens | | | |
| Bicalutamide | 2140242000 | | |
| Flutamide | 2140244000 | | |
| Nilutamide | 2140246000 | | |

| Hormonal therapy | GPI | HCPCS/CPT | ICD |
|---|---|---|---|
| Definitive therapy | GPI | HCPCS | ICD |
| Radical prostatectomy | | 55831, 55840, 55842, 55845, 55866 | ICD-9-PCS<br>6021, 6029, 603, 604, 605, 6061, 6062, 6069<br>ICD-10-PCS<br>0VT00ZZ, 0VT04ZZ, 0VT07ZZ, 0VT08ZZ,<br>0VB00ZZ, 0VB03ZZ, 0VB04ZZ, 0VB07ZZ,<br>0VB08ZZ, 0V500ZZ, 0V503ZZ, 0V504ZZ,<br>0V507ZZ, 0V508ZZ |
| External beam radiation treatment | | <u>CPT</u><br>77401-77416<br><u>HCPCS</u><br>G6003-G6014 | |
| Brachytherapy | | <u>CPT</u><br>7761-77763, 77767-77768, 77770-<br>77772, 77778, 77789, 77750, 77790<br><u>HCPCS</u><br>0394T-0395T | |
| Chemotherapy | GPI | HCPCS | ICD |
| Taxane Chemotherapy | | | |
| Cabazitaxel | 2150000300 | C9276, J9043 | |
| Docetaxel | 2150000500 | J9170, J9171 | |
| Other Chemotherapy | | | |
| Carboplatin | 2110001500 | J9045 | |
| Cisplatin | 2110002000 | J9060, J9062 | |
| Oxaliplatin | 2110002800 | J9263 | |
| Mitoxantrone | 2120005500 | J9293 | |
| Immunotherapy | GPI | HCPCS | ICD |
| Pembrolizumab | 21357953002 | J9271, C9027 | |
| Sipuleucel-T | 2165107000 | Q2043, C9273 | |
| Radium | GPI | HCPCS | ICD |
| Radium-223 | 2160005500 | A9606 | |
| Others | GPI | HCPCS | ICD |
| Lutetium Lu 177 vipivotide tetraxetan<br>Olaparib | 21600045802020<br>21535560 | A9607 | |
| Rucaparib | 21535570 | | |
| Niraparib | 21535550200, | | |

# PFIZER CONFIDENTIAL

| Hormonal therapy | GPI | HCPCS/CPT | ICD |
|---|---|---|---|
| Talazoparib<br>Ketoconazole | 21409902120<br>215355804001<br>1140404000,<br>9630106400,<br>9015404500 | | |
| Radiation therapy | GPI | HCPCS | ICD |
| Brachytherapy | | <u>CPT</u> 7761-77763, 77767-77768, 77770- 77772, 77778, 77789, 77750, 77790 <u>HCPCS</u> 0394T-0395T | |
| External beam radiation treatment | | <u>CPT</u><br>77401-77416<br><u>HCPCS</u><br>G6003-G6014 | |
| Intensity modulated radiation therapy | | G6015-G6016<br><u>CPT:</u> 77385-77386 | |
| Proton beam therapy | | <u>CPT:</u> 77520-77525 | |
| Stereotactic body radiation therapy | | <u>CPT:</u> 77373 | |
| Bone protective agents | GPI | HCPCS | ICD |
| Denosumab | 3004453000 | J0897, C9272 | |
| Ibandronate | 3004204810 | J1740, C9229 | |
| Zoledronic acid | 3004209000 | J3489, Q2051, J3487, J3488,<br>Q4095 | ICD-9-PCS<br>V58.68<br>ICD-10-PCS<br>Z79.83 |
| Pamidronate disodium | 3004206010 | J2430 | |
| Corticosteroids | GPI | HCPCS | ICD |
| Corticosteroids | 22, 8910, 8915 | C9256, J0702, J0704, J1020, J1030, J1040, J1094, J1100, J1700, J1710, J1720, J2650, J2920, J2930, J3300, J3301, J3302, J3303, J7312, J7506, J7509, J7510, J7512, J8540 | |
| Pain medications (analgesics) | | | |
| Non-narcotics | 64 | | |

| Hormonal therapy | GPI | HCPCS/CPT | ICD |
|-------------------------------|-----|-----------|-----|
| Opioids | 65 | | |
| Anti-inflammatory medications | 66 | | |

# **Appendix Table 2. Diagnosis Codes for Comorbidities**

| <b>Conditions and comorbidities</b> | ICD-9-CM | ICD-10-CM |
|---|---|---|
| Charlson comorbidity index (CCI) <sup>1</sup> | | |
| HIV/AIDS | 042–044 | B20–B22, B24 |
| Cerebrovascular disease | 362.34, 430–438 | G45, G46, H34.0, I60–I69 |
| Chronic pulmonary disease | 416.8, 416.9, 490–505, 506.4, 508.1, 508.8 | I27.8, I27.9, J40–J47, J60–J67, J68.4, J70.1, J70.3 |
| Congestive heart failure | 398.91, 402.01, 402.11,<br>402.91, 404.01, 404.03,<br>404.11, 404.13, 404.91,<br>404.93, 425.4–425.9, 428 | I09.9, I11.0, I13.0, I13.2, I25.5, I42.0, I42.5–I42.9, I43, I50, P29.0 |
| Dementia | 290, 294.1, 331.2 | F00–F03, F05.1, G30, G31.1 |
| Diabetes with chronic complication | 250.4–250.7 | E10.2–E10.5, E10.7, E11.2–E11.5, E11.7, E12.2–E12.5, E12.7, E13.2–E13.5, E13.7, E14.2–E14.5, E14.7 |
| Diabetes without chronic complication | 250.0–250.3, 250.8, 250.9 | E10.0, E10.1, E10.6, E10.8, E10.9, E11.0, E11.1, E11.6, E11.8, E11.9, E12.0, E12.1, E12.6, E12.8, E12.9, E13.0, E13.1, E13.6, E13.8, E13.9, E14.0, E14.1, E14.6, E14.8, E14.9 |
| Hemiplegia or paraplegia | 334.1, 342, 343, 344.0–344.6, 344.9 | G04.1, G11.4, G80.1, G80.2, G81, G82, G83.0–G83.4, G83.9 |
| Mild liver disease | 070.22, 070.23, 070.32, 070.33, 070.44, 070.54, 070.6, 070.9, 570, 571, 573.3, 573.4, 573.8, 573.9, V42.7 | B18, K70.0–K70.3, K70.9, K71.3–K71.5, K71.7, K73, K74, K76.0, K76.2–K76.4, K76.8, K76.9, Z94.4 |
| Moderate or severe liver disease | 456.0–456.2, 572.2–572.8 | I85.0, I85.9, I86.4, I98.2, K70.4, K71.1, K72.1, K72.9, K76.5, K76.6, K76.7 |
| Myocardial infarction | 410, 412 | I21, I22, I25.2 |
| Peptic ulcer disease | 531–534 | K25–K28 |
| Peripheral vascular disease | 093.0, 437.3, 440, 441,<br>443.1–443.9, 447.1, 557.1,<br>557.9, V43.4 | I70, I71, I73.1, I73.8, I73.9, I77.1, I79.0, I79.2, K55.1, K55.8, K55.9, Z95.8, Z95.9 |
| Renal disease | 403.01, 403.11, 403.91,<br>404.02, 404.03, 404.12,<br>404.13, 404.92, 404.93, 582,<br>583.0–583.7, 585, 586, 588.0,<br>V42.0, V45.1, V56 | I12.0, I13.1, N03.2–N03.7, N05.2–N05.7, N18, N19, N25.0, Z49.0–Z49.2, Z94.0, Z99.2 |
| Rheumatic disease | 446.5, 710.0–710.4, 714.0–<br>714.2, 714.8, 725 | M05, M06, M31.5, M32–M34, M35.1, M35.3, M36.0 |
| Individual conditions | 262 11 401 vv 405 ···· 427 2 | H25 020 110 112 115 116 167 4 |
| Hypertension Stroke | 362.11, 401.xx-405.xx, 437.2<br>430-434, 436, 362.31-362.34 | H35.039, I10–I13, I15–I16, I67.4<br>I60, I61, I62, I64, I65, I67, H34.1, H34.23, |
| SHORE | 130-131, 130, 302.31-302.3 <del>1</del> | H34.21, H34.0 |
| Acute Coronary Syndrome | 411.x, 410.xx | 124, 121 |
| Angina Pectoris | 413 | 120 |
| Arrhythmia | 427.1, 427.4, 427.41, 427.42,<br>427.5, 427.69, 427.2, 427.60, | I47.0, I47.2, I49.0, I46, I49.3, I49.49, I47.9, I49.40, I49.5, I49.8, I49.9 |

# PFIZER CONFIDENTIAL

| Conditions and comorbidities | ICD-9-CM | ICD-10-CM |
|---|---|---|
| | 427.8, 427.89, 427.9 | |
| Myocardial Infarction | 410, 412 | I21, I22, I25.2 |
| Congestive Heart Failure | 428.xx | 109.9, 111.0, 113.0, 113.2, 125.5, 142.0, |
| | | I42.5-I42.9, I43.x, I50.x, P29.0 |
| Hyperlipidemia | 272.0-272.4 | E78.00, E78.01, E78.1, E78.2, E78.3, |
| | | E78.41, E78.49, E78.5 |
| Low-extremity Arterial | 444.22 | I74.3, I74.4 |
| Occlusive Disease | | |
| Type II Diabetes | 250.0-250.3, 250.7 | E10.0, E10.1, E10.6, E10.8, E10.9, E11.0, |
| | | E11.1, E11.6, E11.8, E11.9, E12.0, E12.1, |
| | | E12.6, E12.8, E12.9, E13.0, E13.1, E13.6, |
| | | E13.8, E13.9, E14.0, E14.1, E14.6, E14.8, |
| | | E14.9 |
| Chronic Obstructive | 490-492, 494, 496 | J40, J41, J42, J43, J47, J44.9 |
| Pulmonary Disease | | |
| Inflammatory bowel disease | | |
| Crohn's disease | 555 | K50 |
| Ulcerative Colitis | 556 | K51 |
| Other cancers | 140-172, 174-184, 186-195, | C00-C43, C45-C60, C62, C63, C67-C76, |
| | 199-209 | C80-C96, C7A, C7B |

**Abbreviations**: HIV: human immunodeficiency virus; ICD-9-CM, International Classification of Diseases, Ninth Revision, Clinical Modification; ICD-10-CM, International Classification of Diseases, Tenth Revision, Clinical Modification

<sup>[1]</sup> Source: Quan, Hude, et al. Coding algorithms for defining comorbidities in ICD-9-CM and ICD-10 administrative data. Medical care (2005): 1130-1139.

# **Document Approval Record**

| Document Name: | C3431052 Non Interventional Protocol - NHTs for mCSPC - VA data a nalyses 06Nov2023 |
|---|---|
| Document Title: | C3431052 Non Interventional Protocol - NHTs for mCSPC - VA data a nalyses 06Nov2023 |

| Signed By: | Date(GMT) | Signing Capacity |
|------------|----------------------|------------------------|
| PPD | 16-Nov-2023 18:36:00 | Business Line Approver |
| PPD | 21-Nov-2023 13:30:23 | Manager Approval |